CLINICAL TRIAL: NCT03636802
Title: Study of the Prevalence, Nature and Contributing Factors of Painful Symptoms of the Musculoskeletal System After Lung Transplantation; Impact on Physical Activity and Quality of Life
Brief Title: Study of the Prevalence of Painful Symptoms of the Musculoskeletal System After Lung Transplantation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-48
Record Dates: First submitted 2018-08-16; First posted 2018-08-17 (Actual); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Respiratory Insufficiency
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- EXPERIMENTAL GROUP: Patient with respiratory failure and on a lung transplant waiting list
  Interventions: Other: Questionnaire BPI

INTERVENTIONS:
Other: Questionnaire BPI — Brief Pain Inventory (BPI) This is a scale of self-assessment, the Concise Pain Questionnaire in French. For all adult patients For any type of pain This is to ask the patient to answer questions in order to learn about us characteristics of his pain (its intensity and its repercussions on the plane biopsychosocial).

SUMMARY:
Pulmonary transplantation (PT) is a therapeutic option now accepted in the management of selected patients who have reached the irreversible and terminal stage of their chronic respiratory insufficiency. Its main indications are: cystic fibrosis and other bronchial diseases, emphysema , interstitial lung diseases with idiopathic pulmonary fibrosis in the foreground, and severe pulmonary hypertension.

The evocation of osteo-articular and musculotendinous pain symptoms in the aftermath of PT is frequent and very diversified. These complications are poorly codified and hinder the rehabilitation and early resumption of physical activity and sports. Few data are available on this subject in the literature.

Following transplantation, improvements in respiratory function, quality of life, and exercise capacity are observed, with large inter-individual variations;

Patients are encouraged to resume physical activity, initially as part of a rehabilitation exercise.

Among the factors limiting exercise, some have been more widely studied, such as muscular deconditioning related to pre-existing chronic respiratory insufficiency , prolonged stay in intensive care, side effects of transplant-related treatments (corticosteroids and immunosuppressants).

Pain is also a factor limiting the recovery of physical activity and quality of life. Pain related directly to thoracotomy surgery has been explored but there is little data available on musculoskeletal pain.

The purpose of this study is to better understand the musculoskeletal pain occurring in the aftermath of a lung transplantation. Conducting this study for a period of 1 year will allow you to move away from the immediate post-transplant time, and the pain associated with the transplant will no longer have any interference.

The main objective of our study is to better know the prevalence of algic manifestations of the musculoskeletal system (osteo-articular, musculotendinous ...) occurring in the year following a TP, and may constitute a brake on the rehabilitation of the musculoskeletal system. effort and recovery of physical activity or sport.

DETAILED DESCRIPTION:
Pulmonary transplantation (PT) is a therapeutic option now accepted in the management of selected patients who have reached the irreversible and terminal stage of their chronic respiratory insufficiency. Its main indications are: cystic fibrosis and other bronchial diseases, emphysema (primary deficit or in the context of COPD), interstitial lung diseases with idiopathic pulmonary fibrosis in the foreground, and severe pulmonary hypertension.

The evocation of osteo-articular and musculotendinous pain symptoms in the aftermath of PT is frequent and very diversified. These complications are poorly codified and hinder the rehabilitation and early resumption of physical activity and sports. Few data are available on this subject in the literature.

Following transplantation, improvements in respiratory function, quality of life, and exercise capacity are observed, with large inter-individual variations.

Patients are encouraged to resume physical activity, initially as part of a rehabilitation exercise.

Among the factors limiting exercise, some have been more widely studied, such as muscular deconditioning related to pre-existing chronic respiratory insufficiency, prolonged stay in intensive care, side effects of transplant-related treatments (corticosteroids and immunosuppressants).

Pain is also a factor limiting the recovery of physical activity and quality of life. Pain related directly to thoracotomy surgery has been explored but there is little data available on musculoskeletal pain.

The purpose of this study is to better understand the musculoskeletal pain occurring in the aftermath of a lung transplantation. Conducting this study for a period of 1 year will allow you to move away from the immediate post-transplant time, and the pain associated with the transplant will no longer have any interference.

The main objective of our study is to better know the prevalence of algic manifestations of the musculoskeletal system (osteo-articular, musculotendinous ...) occurring in the year following a TP, and may constitute a brake on the rehabilitation of the musculoskeletal system. effort and recovery of physical activity or sport.

ELIGIBILITY:
Inclusion Criteria:

Patient over 18

* Having agreed to no opposition
* Registered on the lung transplant waiting list of the CHU de Marseille
* Able to read, understand and complete the self-questionnaires of the study

Exclusion Criteria:

Patient under 18 years

* Patient refusing follow up until 12 months post transplant
* Pregnant women, persons deprived of their liberty, persons under guardianship or trusteeship, persons in an emergency situation
* Person not affiliated to a social security scheme or not entitled to

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient registered on the lung transplant waiting list of the CHU de Marseille
Sampling Method: Non-Probability Sample
Enrollment: 62 (Estimated)
Dates: Start 2018-05-31 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
numbers of patients with symptoms of the musculoskeletal system | 1 years
  numbers of patients presenting symptoms of the musculoskeletal system during the study

CONTACTS AND LOCATIONS:
Overall Officials: EMILIE GARRIDO PRADALIE, Study Director — APHM
Locations (1):
- Assistance Publique Des Hopitaux de Marseille, Marseille, PACA, France